CLINICAL TRIAL: NCT04768959
Title: Cultivating Well-being Beyond Symptomatology in Severe Psychiatric Conditions: A Randomized Controlled Trial
Brief Title: Cultivating Well-being in Severe Psychiatric Conditions
Acronym: FelizMente2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Carmen Valiente Ots, Carmen Valiente Ots, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniversityComplutenseMadrid
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Wellbeing
Keywords: schizophrenia; severe psychiatric conditions; wellbeing; RCT; positive psychology; third-generation psychotherapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: TAU + waiting list (No Intervention): This control group is a waiting list group. Participants received treatment as usual (TAU). Once the RCT is finished, participants have the chance to participate in the intervention group.
- Experimental: TAU + Feliz-Mente Intervention (Experimental): Feliz-Mente (third generation psychotherapy):The intervention is delivered in a group format with a total of 12 sessions and a maximum of 10 patients per group. The protocol consists of specific exercises: 1: welcome and identification of emotions, 2: identification and amplification of positive emotions, 3: regulation of negative emotions, 4: gratitude, 5: forgiveness, 6: self-compassion, 7: personal strengths, 8: loving-kindness and positive interpersonal relationships, 9: values, 10: purpose of life, 11: resilience, 12: keeping the change and farewell party.
  Interventions: Behavioral: FelizMente

INTERVENTIONS:
Behavioral: FelizMente — The intervention aims to improve well-being, without denying the existence of symptoms or problems, focusing on generating positive emotions and actions congruent with the person's values through 11 weekly 90-minute group sessions. The multi-component intervention manual was composed of evidence-based exercises of Positive Psychoterapy Interventions, Acceptance and Commitment Therapy and Mindfulness and was theory driven according the broaden-and-build-theory (Fredrickson, 2001) and the self-serving model of paranoia (Murphy et al., 2018). It was also informed by previous pilot studies carried out on people with paranoid tendencies (see Valiente et al., 2020) and with Severe Psyquiatric Condition samples.
  Other Names: Positive psychotherapy
  Arms: Experimental: TAU + Feliz-Mente Intervention

SUMMARY:
The multicomponet psychological intervention is called Feliz-Mente, with third generation therapy components that aims to improve wellbeing and self-enhancement. Without intervening directly on the symptoms, it is expected to increase positive experiences, the use of personal strengths and positive relationships, and aims to build a more meaningful self-narrative in persons with severe psychiatric conditions. Feliz-Mente is a group intervention of 12 sessions in which participants are expected to perform exercises during and between sessions to improve treatment adherence and daily practice. The design for the present study is a randomized controlled trial, which compares the post-intervention measures of the experimental group (group receiving the intervention) with the post-intervention measures of the control group (treatment as usual + waiting list).

ELIGIBILITY:
Inclusion Criteria:

* 1) were aged 18-65 years
* 2) had a minimum of motivation and commitment to participate in group therapy

Exclusion Criteria:

* 1) limited cognitive resources or serious formal thinking disorder and/or
* 2) a concurrent diagnosis of substance dependence or a severe personality disorder that could interfere with benefiting from a psychotherapy group.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Well-being | Change from Well-being at 12 weeks and 6 months
  Psychological Well-Being Scales (Ryff, 1995)
Well-being | Change from Well-being at 12 weeks and 6 months
  Satisfaction with life Scale ( Diener et al. 1985)

SECONDARY OUTCOMES:
Self-esteem | Change from self-esteem at 12 weeks and 6 months
  Rosenberg self-esteem scale (Rosenberg, 1965)
Attachment | Change from Attachment at 12 weeks and 6 months
  Relationship Questionnaire (Bartholomew and Horowitz, 1991)
Psychological Symptoms | Change from Psychological Symptoms at 12 weeks and 6 months
  Symptom Checklist 90-Revised (SCL-90-R; Derogatis, 2002)
Experiential Avoidance | Change from Experiential Avoidance at 12 weeks and 6 months
  The Acceptance and Action Questionnaire (AAQ; Hayes et al.,2004)

CONTACTS AND LOCATIONS:
Locations (1):
- Carmen Valiente, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code